CLINICAL TRIAL: NCT03609554
Title: Improvement in Adolescents With a History of Back Pain After Pilates
Brief Title: Improvements in Adolescents With Back Pain After Pilates
Acronym: PilatesBack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Noelia González-Gálvez, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NGonzalez-Galvez
Record Dates: First submitted 2018-07-04; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Back Pain
Keywords: trunk flexor endurance; trunk extensor endurance; hamstring extensibility
MeSH Terms: conditions — Back Pain | interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates (Experimental): The Pilates exercise programme was implemented over 6 weeks, with 2 sessions/week (55 minutes/session).
  Interventions: Other: Pilates
- Control (No Intervention): Adolescents assigned to the CG did not receive any structured exercise programme; they just attended their usual Physical Education sessions.

INTERVENTIONS:
Other: Pilates — The Pilates exercise programme was implemented over 6 weeks, with 2 sessions/week (55 minutes/session). The Pilates programme was conducted by the Physical Education teacher, who was certified in Pilates training. The Pilates programme began at the basic level, incorporating more difficult principles and exercises gradually. The sessions were divided into the warm-up (7 min), the main part (41 min), and the cool down (7 min). Tt concentrated on basic Pilates exercises involving the principal regions of the body (spine flexions, extensions and rotations; hip flexions, extensions and rotations; and shoulder abductions, adductions and rotations).
  Arms: Pilates

SUMMARY:
The main physical condition factor related to back pain and mobility among adolescents are trunk endurance and hamstring extensibility. The Pilates Method (PM) can be used as a specific exercise technique to train trunk endurance and hamstring extensibility, but there is little evidence regarding its effect in adolescents with a history of back pain. The objective of this study is to determine whether Pilates is effective for improving the trunk endurance and hamstring extensibility of adolescents with a history of back pain and to determine the differences between the sexes. The sample was composed of 52 students with a mean age of 14.44 ± 0.7 years who had suffered back pain during the past year. They were distributed into the Pilates Exercise Group (PEG, n = 26) and the Control Group (CG, n = 26). The Pilates programme was conducted over 6 weeks. For measuring trunk flexion and extension endurance, the bench trunk curl (BTC) test and the Sorensen (SOR) test were used, respectively. Hamstring extensibility was measured with the toe touch (TT) test. After the Pilates intervention, either the whole sample or males and females separately improved significantly (p ≤ 0.05) in the BTC, SOR or TT test.

DETAILED DESCRIPTION:
Back pain during the adolescent years is a precursor to chronic back pain in adulthood. The prevalence of back pain among schoolchildren is growing across the world, and it is similar to that of the adult population. Back pain is the first cause of disability in the world.

The main physical condition factor related to back pain and mobility among adolescents are trunk endurance and hamstring extensibility. The Pilates Method (PM) can be used as a specific exercise technique to train trunk endurance and hamstring extensibility, but there is little evidence regarding its effect in adolescents with a history of back pain.

The objectives of this study was: a) to analyse the effect of a Pilates programme on trunk endurance and extensibility in adolescents with a history of back pain and b) to determine the differences between the sexes.

The present research was a 6-week randomised controlled trial in which adolescents with a history of back pain were randomly assigned to a Pilates-based exercise group (PEG; n = 26) and a control group (CG; n = 26).

The sample was composed of 52 students with a mean age of 14.44 ± 0.7 years who had suffered back pain during the past year. They were distributed into the Pilates Exercise Group (PEG, n = 26) and the Control Group (CG, n = 26).

The Pilates exercise programme was implemented over 6 weeks, with 2 sessions/week (55 minutes/session). Adolescents assigned to the CG did not receive any structured exercise programme; they just attended their usual Physical Education sessions.

The Pilates programme was conducted by the Physical Education teacher, who was certified in Pilates training. The Pilates programme began at the basic level, incorporating more difficult principles and exercises gradually.

For measuring trunk flexion and extension endurance, the bench trunk curl (BTC) test and the Sorensen (SOR) test were used, respectively. Hamstring extensibility was measured with the toe touch (TT) test. After the Pilates intervention, either the whole sample or males and females separately improved significantly (p ≤ 0.05) in the BTC, SOR or TT test.

ELIGIBILITY:
Inclusion Criteria:

* having had a history of back pain last year
* being physically active in school physical education sessions

Exclusion Criteria:

* presenting any musculoskeletal, neurological, cardiological, metabolic or rheumatic alteration
* missing more than one session of the programme (91.66% attendance)

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2016-01-16 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
Trunk flexor endurance | Pre and Post-intervention: change after 6 weeks of intervention
  The bench trunk curl (BTC) test was used to evaluate trunk flexor endurance. The result is register in repetitions numbers. Higher values represent a better outcome.
Isometric trunk extension | Pre and Post-intervention: change after 6 weeks of intervention
  Isometric trunk extension endurance was measured using the Sorensen (SOR) test. The result is register in seconds. Higher values represent a better outcome.
Hamstring extensibility | Pre and Post-intervention: change after 6 weeks of intervention
  The toe touch (TT) test was used to evaluate hamstring extensibility. The result is register in centimeters. Higher values represent a better outcome.

SECONDARY OUTCOMES:
Weight | Pre and Post-intervention: change after 6 weeks of intervention
  Weight was measured using a SECA 762 scale (SECA, Germany) in kilograms.
Height | Pre and Post-intervention: change after 6 weeks of intervention
  Height was measured using a GPM anthropometer (Siber-Hegner, Switzerland) in meters.

CONTACTS AND LOCATIONS:
Overall Officials: Noelia González, PhD., Principal Investigator — UCAM

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peterson L, Haladay DE. Pilates-based exercise in the treatment of a patient with persistent low back pain following transforaminal lumbar interbody fusion. Physiother Theory Pract. 2020 Apr;36(4):542-549. doi: 10.1080/09593985.2018.1488905. Epub 2018 Jun 26. PMID 29944036
- [Background] Cruz-Diaz D, Romeu M, Velasco-Gonzalez C, Martinez-Amat A, Hita-Contreras F. The effectiveness of 12 weeks of Pilates intervention on disability, pain and kinesiophobia in patients with chronic low back pain: a randomized controlled trial. Clin Rehabil. 2018 Sep;32(9):1249-1257. doi: 10.1177/0269215518768393. Epub 2018 Apr 13. PMID 29651872
- [Background] Miyamoto GC, Franco KFM, van Dongen JM, Franco YRDS, de Oliveira NTB, Amaral DDV, Branco ANC, da Silva ML, van Tulder MW, Cabral CMN. Different doses of Pilates-based exercise therapy for chronic low back pain: a randomised controlled trial with economic evaluation. Br J Sports Med. 2018 Jul;52(13):859-868. doi: 10.1136/bjsports-2017-098825. Epub 2018 Mar 10. PMID 29525763
- [Background] Vaquero-Cristobal R, Lopez-Minarro PA, Alacid Carceles F, Esparza-Ros F. [THE EFFECTS OF THE PILATES METHOD ON HAMSTRING EXTENSIBILITY, PELVIC TILT AND TRUNK FLEXION]. Nutr Hosp. 2015 Nov 1;32(5):1967-86. doi: 10.3305/nh.2015.32.5.9678. Spanish. PMID 26545650
- [Background] Kibar S, Yardimci FO, Evcik D, Ay S, Alhan A, Manco M, Ergin ES. Can a pilates exercise program be effective on balance, flexibility and muscle endurance? A randomized controlled trial. J Sports Med Phys Fitness. 2016 Oct;56(10):1139-1146. Epub 2015 Oct 16. PMID 26473443
- [Background] Miranda IF, Souza C, Schneider AT, Chagas LC, Loss JF. Comparison of low back mobility and stability exercises from Pilates in non-specific low back pain: A study protocol of a randomized controlled trial. Complement Ther Clin Pract. 2018 May;31:360-368. doi: 10.1016/j.ctcp.2017.12.005. Epub 2017 Dec 8. PMID 29248397